CLINICAL TRIAL: NCT03900039
Title: Randomized Control Trial of Four Bearing Surfaces in Primary Total Hip Arthroplasty in Patients Over the Age of 18 Years
Brief Title: An Assessment of 4 Different Bearing Types in Hip Replacement Types to Analsye the Lowest Wear Rates of Polyethylene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: #04-025
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Arthroplasty Complications; Hip Arthritis
Keywords: Hip arthroplasty; Tribology; wear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessment of the implants was done by a secondary center that was unaware of which the bearing type was in which patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Conventional Polyethylene versus metal head (Active Comparator): This is the more conventional group bearing surfaces
  Interventions: Device: Highly Cross Linked Polyethylene and oxidized zirconium femoral head
- Conventional Polyethylene versus oxidized zirconium head (Experimental): This group uses the more conventional polyethylene against the newer head
  Interventions: Device: Highly Cross Linked Polyethylene and oxidized zirconium femoral head
- Newer Cross linked Polyethylene metal head (Experimental): In this group we continued with the conventional polyethylene, but added in the new type of head (oxidized zirconium)
  Interventions: Device: Highly Cross Linked Polyethylene and oxidized zirconium femoral head
- Newer Cross linked Polyethylene versus oxidized zirconium head (Experimental): In this group, we added both the new head and the new polyethylene
  Interventions: Device: Highly Cross Linked Polyethylene and oxidized zirconium femoral head

INTERVENTIONS:
Device: Highly Cross Linked Polyethylene and oxidized zirconium femoral head — Differing bearing surfaces:
  1. Conventional polyethylene versus cobalt Chrome heads
  2. Conventional polyethylene versus Oxidized Zirconium heads
  3. Highly Cross-linked polyethylene versus Cobalt Chrome heads
  4. Highly Cross-linked polyethylene versus Oxidized Zirconium heads
  Other Names: Varilast - from Smith & Nephew

SUMMARY:
The aim of the study is to assess the ideal bearing surfaces in hip replacement by comparing 4 different combinations. In a hip replacement this means what the head and the socket liner are made of.

DETAILED DESCRIPTION:
In hip replacements, arguably the most important thing for survivorship is what rubs against what.

Traditionally surgeons used metal (Cobalt-Chrome) against a conventional polyethylene (plastic). More recently (around 15 years ago) a newer more dense type of polyethylene (called XLPE) had been developed and a new type of head called Oxidized Zirconium was also developed.

In this trial, adults who were undergoing hip replacements were randomized assigned into one of the four groups:

Group 1: old plastic vs metal head Group 2: Old plastic against Oxidized Zirconium Group 3: New plastic versus metal head Group 4 New plastic vs Oxidized Zirconium

All patients were followed up for a minimum of 10 years to assess which group wore the most amount of polyethylene and which group had the best survival rate.

ELIGIBILITY:
Inclusion Criteria:

* All adults with no history of cancer, infection of the hip and with the capacity to make informed consent for the trial

Exclusion Criteria:

* those under the age of 18 and over 65. Those with a history of cancer and infection. Those without the capacity to make an informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-07-26 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Wear rates of polyethylene over 10 years | Over 10 years of wear rates
  Linear and volumetric wear were measured in the most recent radiographs using a computer software package (Polyware Rev. 5; Draftware).

SECONDARY OUTCOMES:
Survivorship of implant combinations | over 10 years
  Assess linear and volumetric wear to assess if those bearing surfaces require to be revised (exchanged) during the experimental period in one group more than the others

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atrey A, Ward SE, Khoshbin A, Hussain N, Bogoch E, Schemitsch EH, Waddell JP. Ten-year follow-up study of three alternative bearing surfaces used in total hip arthroplasty in young patients: a prospective randomised controlled trial. Bone Joint J. 2017 Dec;99-B(12):1590-1595. doi: 10.1302/0301-620X.99B12.BJJ-2017-0353.R1. PMID 29212681
- [Result] Rames RD, Stambough JB, Pashos GE, Maloney WJ, Martell JM, Clohisy JC. Fifteen-Year Results of Total Hip Arthroplasty With Cobalt-Chromium Femoral Heads on Highly Cross-Linked Polyethylene in Patients 50 Years and Less. J Arthroplasty. 2019 Jun;34(6):1143-1149. doi: 10.1016/j.arth.2019.01.071. Epub 2019 Feb 5. PMID 30808529